CLINICAL TRIAL: NCT05636670
Title: Assessment of Cognitive Function and Gut Microbiota Analysis in Real World Patients With Lupus Cerebrovascular Disease: a Retrospective and Prospective Cohort Study
Brief Title: Assessment of Cognitive Function and Gut Microbiota Analysis in Real World Patients With Lupus Cerebrovascular Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: NFEC-2022-417
Record Dates: First submitted 2022-11-13; First posted 2022-12-05 (Actual); Last update posted 2022-12-05 (Actual); Status verified 2022-11

CONDITIONS: Lupus Erythematosus, Systemic; Gastrointestinal Microbiome
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples Without DNA — serum and stool specimens
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- SLE group: 1. The researcher signed the informed consent voluntarily;
  2. Male or female patients aged 14-55 years;
  3. Patients diagnosed with systemic lupus erythematosus are classified according to the European League against Rheumatism (EULAR)/American College of Rheumatology (ACR) joint classification criteria for SLE in 2019.
  4. Patients who need to undergo head imaging examination according to the judgment of treating doctors, and the results of head imaging examination are not consistent with changes in cerebrovascular disease.
  5. no antibiotics have been taken in the past 2 weeks;
- NPSLE epilepsy group: 1. The researcher signed the informed consent voluntarily;
  2. Male or female patients aged 14-55 years
  3. Patients diagnosed with systemic lupus erythematosus are classified according to the European League against Rheumatism (EULAR)/American College of Rheumatology (ACR) joint classification criteria for SLE in 2019.
  4. Patients who need MRI according to the judgment of the treating doctor, and reveal that the MRI suggests cerebrovascular disease;
  5. no antibiotics have been taken in the past 2 weeks;
- Healthy control group: 1. Male or female patient volunteers aged 14-55 from the Health Examination Center of Nanfang Hospital,
  2. Voluntary signing of informed consent;
  3. no systemic disease;
  4. According to the judgment of the researchers, healthy volunteers matching SLE group in age, gender and education level were selected as the control group;

SUMMARY:
Based on clinical manifestations, laboratory data and intestinal microflora detection, the cognitive function characteristics of patients with systemic lupus erythematosus and cerebrovascular disease and its relationship with intestinal microflora were analyzed to explore the possible pathogenesis of lupus cerebrovascular disease.

DETAILED DESCRIPTION:
This study was a retrospective and prospective cohort study. They were divided into three groups, namely SLE group, SLE cerebrovascular disease group and healthy control group. Each group included 60 patients [Anticipated].

1. Retrospective study: The SLE patients admitted to Nanfang Hospital from 2018 to 2022 were retrieved. The patients enrolled from September 2018 to September 2021 applied for exemption from informed consent, and the patients enrolled from September 2021 to September 2022 voluntarily signed informed consent. Patients were selected according to inclusion and exclusion criteria, and clinical and laboratory data of all subjects were recorded.
2. Prospective study: Obtain the consent of the subjects, sign the informed consent, and record the clinical and laboratory examination data of all the subjects.

(1) Cognitive function assessment; (2) Fresh stool and serum were collected, and 16s rRNA technology was used for intestinal flora detection, and QIIME2 platform was used for flora analysis; Serum inflammatory factors were detected and metabolomic analysis was performed.

The clinical data of all enrolled patients were statistically analyzed.

ELIGIBILITY:
Inclusion Criteria:

Retrospective study

* Patients enrolled from September 2018 to September 2021 applied for exemption from informed consent, and patients enrolled from September 2021 to September 2022 signed informed consent voluntarily.
* Male or female patients aged 14-55 years;
* Patients diagnosed with systemic lupus erythematosus are classified according to the European League against Rheumatism (EULAR)/American College of Rheumatology (ACR) joint classification criteria for SLE in 2019.
* Cranial imaging examination was performed, and the results of cranial imaging examination were consistent with cerebrovascular disease changes.

Prospective Research:

SLE group:

* The researcher signed the informed consent voluntarily;
* Male or female patients aged 14-55 years;
* Patients diagnosed with systemic lupus erythematosus are classified according to the European League against Rheumatism (EULAR)/American College of Rheumatology (ACR) joint classification criteria for SLE in 2019.
* Patients who need to undergo head imaging examination according to the judgment of treating doctors, and the results of head imaging examination are not consistent with changes in cerebrovascular disease.
* No antibiotics have been taken in the past 2 weeks; SLE cerebrovascular disease group
* The researcher signed the informed consent voluntarily;
* Male or female patients aged 14-55 years
* Patients diagnosed with systemic lupus erythematosus are classified according to the European League against Rheumatism (EULAR)/American College of Rheumatology (ACR) joint classification criteria for SLE in 2019.
* no antibiotics have been taken in the past 2 weeks;

Healthy control group:

* Male or female patient volunteers aged 14-55 from the Health Examination Center of Nanfang Hospital,
* Voluntary signing of informed consent;
* No systemic disease;
* According to the judgment of the researchers, healthy volunteers matching SLE group in age, gender and education level were selected as the control group;

Exclusion Criteria:

* Patients with other autoimmune diseases;
* Brain imaging suggested central nervous system infection, space occupation and other manifestations.
* Patients with malignant tumors and active tuberculosis;
* Pregnancy, lactation or intended pregnancy, women of childbearing age do not use effective contraceptive measures (IUD, oral contraceptives and obstruction measures);
* History of cerebrovascular disease not associated with SLE as determined by the investigator
* The researcher judged that it is not suitable to participate in this researcher.

Ages: 14 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Diagnostic criteria: Patients diagnosed with systemic lupus erythematosus are classified as SLE by the European League against Rheumatism (EULAR)/American College of Rheumatology (ACR) 2019.
  Brain imaging cerebrovascular changes were defined as: great vascular lesions including cerebral infarction, cerebral hemorrhage, venous sinus thrombosis; Microvascular lesions include leukodystrophy, cerebral atrophy, perivascular space enlargement, lacunar infarction, cerebral microhemorrhage focus, and recent subcortical infarction.
Sampling Method: Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-09-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Assess changes in cognitive function by Mini-mental State Examination | Baseline, months 3, 6
  Score on a scale of 27-30: normal; Score<27 points: cognitive dysfunction; 21-26, mild; 10-20, moderate 0-9; Severe
Assess changes in cognitive function by Montreal Cognitive Assessment | Baseline, months 3, 6
  The total score of the scale is 30 points, and the test results show a normal value of ≥26 points.
Assess changes in anxiety by Self-Rating Anxiety Assess changes in anxiety by Self-Rating Anxiety Scale | Baseline, months 3, 6,
  The cut-off value of the SAS standard score is 50 points, of which 50-59 is mild anxiety, 60-69 is moderate anxiety, and 70 points or more is severe anxiety.
Assess depressive mood changes by Self-rating depression scale Assess depressive mood changes by Self-rating depression scale 8/5000 Assess depressive mood changes by Self-rating depression scale | Baseline, months 3, 6
  The dividing value of the SDS standard score is 53 points, with 53-62 being mild depression, 63-72 being moderate depression, and 73 points or more being severe depression.
Assess changes in memory and executive ability by memory and executive screening | Baseline, months 3, 6
  Out of 100, the memory factor is 50, and the execution factor is 50. The 3 indicators of MES (memory score, execution score, and total score) correlated significantly with age, with older age scoring lower and no significant correlation with educational attainment.
Assess changes in cognitive function by auditory verbal learning test | Baseline, months 3, 6
  -1.5SD (50-59 years: 4 points; 60-69 years old: 3 points; 70-89: 2 points); -1.0SD (50-59 years: 5 points; 60-69 years old: 4 points; 70-89:3 points)
Assess changes in cognitive function by Rey-Osterrieth complex figure | Baseline, months 3, 6,
  The total score is 36 points, and the lower the score, the worse it gets
Assess changes in cognitive function by verbal fluency test | Baseline, months 3, 6,
  1 point is awarded for each correct one, and the number of correctly enumerated within 1 minute is the total score. ≥11 points are normal.
Assess changes in cognitive function by shape trails test | Baseline, months 3, 6
  Record the total number of elapsed and first-minute arrivals as well as the number of prompts one
Assess changes in cognitive function by StroopColor-WordTest | Baseline, months 3, 6,
  The amount of interference reflected includes: SIE time consumption = card C - card B time consumed: SIE correct number = card B - card C correct number, the larger the SIE indicates that the more severe the impairment of executive function.
Assess changes in cognitive function by Clock Drawing Test | Baseline, months 3, 6,
  The total score is 30 points, CDT30-A is 4 out of 4, and ≤ 2 points are cognitive impairment; CDT30-B scored 26 out of 26, with ≤17 being rated as impaired cognitive function
Assess changes in cognitive function by digit span test | Baseline, months 3, 6
  Each correct answer is counted as 1 point for a string of numbers, and the total score = smooth back + reverse recitation.
Assess changes in cognitive function by symbol digit modalities test | Baseline, months 3, 6
  The number of correctly filled in within 90s is the final score.
Assess changes in cognitive function by functional activities questionnaire | Baseline, months 3, 6
  The total score is 30 points. A score of > 9 indicates social activity dysfunction.
Assess quality of life changes by Activity of Daily Living Scale | Baseline, months 3, 6
  The total score is 80 points, the higher the score, the more impaired the ability to live a daily life
Assess changes in sleep quality by Pittsburgh sleep quality index | Baseline, months 3, 6
  The total score ranges from 0~21, and the higher the score, the worse the sleep quality.
Changes in the intestinal flora | Baseline, months 3, 6
  Intestinal microbiota detection using 16s rRNA technology

CONTACTS AND LOCATIONS:
Overall Officials: Qin Huang, MD, Study Director — Southern Medical University
Locations (1):
- Qin Huang, Guangzhou, Guangdong, China